CLINICAL TRIAL: NCT02354742
Title: Echocardiography-Guided Resuscitation in Severe Sepsis and Septic Shock Vs. Early Goal-Directed Therapy: Pilot Study
Brief Title: Echo vs. EGDT in Severe Sepsis and Septic Shock
Acronym: ECHO RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1024925
Record Dates: First submitted 2014-11-03; First posted 2015-02-03 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Echocardiography; EGDT; Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Goal Directed Therapy (EGDT) (Active Comparator): EGDT is currently standard of care in management of septic shock, so assignment to this treatment arm will confer no additional risk above that of standard of care. EGDT utilizes placement of a central venous catheter, an arterial catheter, and administration of intravenous fluid and vasoactive medications. EGDT uses central venous catheter to assess central venous pressure and ScVO2.
  Interventions: Other: EGDT fluid resuscitation
- Echo Guided Fluid Resuscitation (Experimental): The echo arm also utilizes placement of a central venous catheter, an arterial catheter, and administration of intravenous fluid and vasoactive medications, all of which are interventions found in standard care. The central venous pressure will not be monitored in this arm. Instead, decisions for giving fluids will be directed by the results of Echocardiography. Echocardiography poses no known risk to the patient, and it is non-invasive. The only risk of echocardiography is that of misdiagnosis.
  Interventions: Other: Echo guided fluid resuscitation

INTERVENTIONS:
Other: Echo guided fluid resuscitation — Patients will have their fluid resuscitation care guided by measurements obtained during an echo.
  Arms: Echo Guided Fluid Resuscitation
Other: EGDT fluid resuscitation — Patients will have their fluid resuscitation care guided by an EGDT protocol, which is currently used as standard of care.
  Arms: Early Goal Directed Therapy (EGDT)

SUMMARY:
Echocardiography (cardiac ultrasound) is being used more often in the critical care setting for management of severe infection (septic shock). Early studies show echocardiography to be useful in these patients, but at this time, there are no good clinical trials to justify its use.

Our study goals/objectives are as follows:

1. To conduct an unblinded, two-group randomized controlled clinical trial to compare an echocardiography-guided resuscitation protocol with an Early Goal Directed Therapy (EGDT) protocol in patients with severe sepsis or septic shock.
2. Demonstrate that a sepsis treatment protocol using transthoracic echocardiography and other non-invasive assessments of cardiac output will result in more rapid resolution of septic shock compared to invasive EGDT.
3. Demonstrate patients receiving the non-invasive echocardiography protocol will receive less administration of intravenous fluid.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Suspected infection
* Two or more systemic inflammatory response syndrome (SIRS) criteria

  * White blood cell count less than 4,000 per mm3, greater than 12,000 per mm3, or differential with greater than 10% immature forms
  * Heart rate greater than 90 beats per minute
  * Respiratory rate greater than 20 breaths per minute or paCO2 less than 32 mmHg
  * Temperature less than 36°C or greater than 38°C
* Evidence of refractory hypoperfusion attributed to sepsis (one or more of the following):

  * Systolic blood pressure less than 90 mmHg despite an intravenous fluid challenge of at least 30ml/kg (a portion of this may be albumin equivalent)
  * Blood lactate level at least 4 mmol/L.
* Intention to place an arterial catheter.
* Intention to place a central venous catheter.

Exclusion criteria:

* Known pregnancy
* Requirement for immediate surgery
* Hypotension attributed to alternative cause
* Treating physician deems the patient is moribund
* Treating physician deems aggressive care is unsuitable
* Contraindication to central venous catheterization or arterial catheterization
* Advanced directives restricting implementation of the protocol
* Significant pathology of the chest or abdominal wall that would make transthoracic echocardiography impossible (burns, chest trauma, etc.)
* Children under the age of 18 will not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Serial organ failure assessment (SOFA) scores in both treatment arms | up to 72 hours

SECONDARY OUTCOMES:
Inpatient mortality in both treatment arms | Up to ~7 days (Occurring during hospital stay).
Time to lactate clearance in both treatment arms | Up to ~7 days (Occurring during ICU hospital stay).
Number of ICU-Free days | 28 days
Daily and cumulative fluid balance in both treatment arms | Up to ~7 days (Occurring during ICU hospital stay).
Number of ventilator-free days | Up to ~7 days (Occurring during ICU hospital stay).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lanspa, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lanspa MJ, Burk RE, Wilson EL, Hirshberg EL, Grissom CK, Brown SM. Echocardiogram-guided resuscitation versus early goal-directed therapy in the treatment of septic shock: a randomized, controlled, feasibility trial. J Intensive Care. 2018 Aug 13;6:50. doi: 10.1186/s40560-018-0319-3. eCollection 2018. PMID 30123511